CLINICAL TRIAL: NCT03506945
Title: Mobile Web-based Behavioral Intervention for Improving Caregiver Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brent Mausbach, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180454; R01AG061941 (NIH)
Record Dates: First submitted 2018-04-06; First posted 2018-04-24 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Depressive Symptoms; Stress, Psychological
MeSH Terms: conditions — Depression; Stress, Psychological | interventions — Bibliotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPEP (Experimental): Behavioral Activation Therapy - Increase engagement in pleasant activities as a mechanism for reducing distress and improving overall well-being. Participants will use an online web tool to select and schedule activities they deem will be rewarding and fulfilling. They will then track their engagement in these activities on a weekly basis.
  Interventions: Behavioral: mPEP
- Bibliotherapy (Active Comparator): Bibliotherapy - Develop improved coping and problem-solving skills. Participants will receive bibliotherapy handouts describing various means of managing their distress and solving caregiving-related problems.
  Interventions: Behavioral: Bibliotherapy

INTERVENTIONS:
Behavioral: mPEP — Behavioral Activation Therapy
  Arms: mPEP
Behavioral: Bibliotherapy — Provide educational material on coping strategies pertinent to caregivers
  Arms: Bibliotherapy

SUMMARY:
Caregivers suffer great amounts of distress that significantly impacts their mental and physical well-being, yet caregivers' access to quality, evidence-based care is currently very limited. The public health significance of the proposed study is that our internet and mobile-based web intervention will (1) significantly reduce caregiver distress and improve caregivers' overall well-being, and (2) dramatically increase caregivers' access to high quality, evidence-based care at relatively low cost.

DETAILED DESCRIPTION:
Over 15 million men and women provide informal caregiving services to family members who have dementia. The literature is replete with evidence that caregiving results in high rates of depression and distress, and potentially high rates of physical morbidity. For example, 40% of caregivers are at risk for depression compared to just 5% of non-caregiving older adults. Further, increased symptoms of depression and distress in caregivers are associated with accelerated risk for developing cardiovascular disease. Thus, efficacious interventions for reducing caregiver distress appear potentially valuable for both mental and physical well-being.

Given the distress experienced by caregivers, it is no surprise that over 80 intervention studies for reducing caregiver distress have been published. The message from these studies is that caregiver interventions, in general, are effective for reducing distress. Yet, the implementation of Evidence Based Treatments (EBTs) continues to be a challenge. Despite identification of EBTs, their use at the community-level has been absent. In 2007, NIH sponsored a workshop on the use of EBTs for caregivers. The conclusion was that "The majority of effective interventions for caregivers were not being implemented through the aging network." Ten years later, this lack of implementation remains. It is critical that scientists develop interventions for caregivers with maximal reach and minimal cost. Currently, most caregiver intervention frameworks require caregivers to meet with a therapist in one of four formats: a) face-to-face meetings with a therapist outside the caregiver's home, b) face-to-face meetings with a therapist in the caregiver's home, c) in-person, group-based meetings, or d) phone-based interventions in which caregivers call a therapist or support group. While possibly efficacious, these therapeutic formats are limited because: a) community agencies serving caregivers do not offer EBTs, b) the interventions are often not accessible to caregivers who reside outside the care network, c) they require caregivers to attend therapy sessions on specific days and times that may not be convenient for them, or d) they may require caregivers to find alternate care for their care recipients while they attend the therapy. To address these limitations, the investigators have adapted an evidence-based, brief Behavioral Activation (BA) program to be delivered to caregivers via mobile phones with internet-based capabilities, thereby increasing caregivers' access to quality care. This mobile intervention is now being tested in this full-scale trial. The investigators will test mechanisms of action, namely that increased behavioral activation promotes well-being in caregivers. To do so, the investigators will recruit and randomize 200 caregivers to receive either a mobile BA intervention (N = 100) known as the mobile pleasant events program (mPEP), or a web-based bibliotherapy condition (N = 100) teaching skills on coping with caregiving. Participants will be assessed for depressive symptoms, positive and negative affect, well-being, and blood pressure at baseline, 3-months, 9-months, and 15-months follow-up time points.

ELIGIBILITY:
Inclusion Criteria -

* English-speaking
* Spouse or Child Caregiver of a loved-one with Alzheimer's Disease or Related Dementia (ADRD)
* Aged 40 years or older at the time of enrollment
* Providing at least 20 hours of in-home care per week
* Screening positive for mild depressive symptoms (CESD-R≥16).

Exclusion Criteria -

* Diagnosed with a terminal illness
* Demonstrates cognitive impairment (MMSE<27)
* Severe hypertension (>200/120 mm Hg)
* Participating in another active caregiver intervention (other than support groups)
* Receiving psychiatric care for serious mental illnesses such as schizophrenia or bipolar disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent T Mausbach, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers. The PI will determine who is authorized to have copies of what types of data and when the data will be available. Publicizing availability of the data after main results from the study have been published, and providing a USB or CD containing the data to individuals who express interest, will ensure that maximum data sharing occurs. We will make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to use the data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate computer technology; and (3) a commitment to destroy or return the data after analyses are completed.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months of close of the trial
Access Criteria: The PI will determine who is authorized to have copies of what types of data and when the data will be available. Publicizing availability of the data after main results from the study have been published, and providing a USB or CD containing the data to individuals who express interest, will ensure that maximum data sharing occurs.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment centered on community providers and research organizations serving caregivers and persons with dementia, as well as community-based caregiver support groups. Further recruitment occurred via digital and print advertisement.
Groups:
- Mobile Pleasant Events Program (mPEP): This arm consists of 12 weeks of behavioral activation therapy delivered via smart phone or smart device (e.g., iPAD).
- Psychoeducation: This arm consists of 12 weeks of digital psychoeducation consisting of a comprehensive resource guide containing materials on coping with specific caregiver stresses (e.g., developing problem-solving skills; managing care receiver problem behaviors; improving communication).
Period: Overall Study
Arm/Group | Mobile Pleasant Events Program (mPEP) | Psychoeducation
Started | 93 | 91
Completed | 63 | 52
Not Completed | 30 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Pleasant Events Program (mPEP) | Psychoeducation | Total
Number analyzed (Participants) | 93 | 91 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (11.3) | 63.1 (11.2) | 63.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 82 | 162
  Male | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 65 | 71 | 136
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 16 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 72 | 70 | 142
  Unknown or Not Reported | 16 | 9 | 25
Center For Epidemiologic Studies Depression Scale - Revised (CESD-R) [Mean (Standard Deviation); unit: Scores on a Scale] — Scale consists of 20 questions with individual item responses ranging from 0-4 (total range for scale is 0-80, with higher score indicating greater depression)
  Scores on a Scale | 19.7 (13.7) | 19.0 (13.2) | 19.4 (13.4)
Positive Affect [Mean (Standard Deviation); unit: Scores on a Scale] — Positive and Negative Affect Scale (PANAS) - Positive Affect Score. Scale consists of 10 items, individual items rated from 1-5 (total range for scale = 10-50, with higher score indicating greater positive affect)
  Scores on a Scale | 28.4 (7.1) | 28.4 (6.3) | 28.4 (6.7)
Negative Affect [Mean (Standard Deviation); unit: Scores on a Scale] — Positive and Negative Affect Scale (PANAS) - Negative Affect Score. Scale consists of 10 items, individual items rated from 1-5 (total range for scale = 10-50, with higher score indicating greater negative affect.
  Scores on a Scale | 22.7 (7.5) | 22.1 (6.4) | 22.4 (7.0)
Quality of Life [Mean (Standard Deviation); unit: Scores on a Scale] — Dementia Quality of Life Scale for Older Family Carers (DQoLOC). Scale consists of 22 items, each item is rated from 1-5. The total range for the scale is 22-110, with higher score indicating greater quality of life.
  Scores on a Scale | 60.2 (12.4) | 60.3 (11.9) | 60.2 (12.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 124.8 (17.8) | 122.4 (17.8) | 123.7 (17.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.9 (7.8) | 75.8 (10.1) | 77.4 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies Depression Scale--Revised (CESD-R)
Description: 20 item scale measuring Depressive Symptoms. Each item rated on a range of 0-4 and items are summed to create a total score (Range = 0-80). Higher scores denote greater depressive symptoms.
Time Frame: 15-months
Population: Participants in each group dropped out or were lost to follow-up
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | mPEP | Bibliotherapy
Number analyzed (Participants) | 63 | 52
Score on a scale | 16.9 (1.6) | 14.9 (1.8)

2. Secondary Outcome: Positive and Negative Affect Scale (PANAS)
Description: Positive and Negative Affect Scale (PANAS). There are 10 items asking about Positive Affect, each item is rated on a range of 1-5. All 10 items are summed to create a total score (Range = 10-50) There are 10 items asking about Negative Affect, each item is rated from 1-5, and items are summed to create an overall score (Range = 10-50). Higher scores denote greater positive and negative affect, respectively.
Time Frame: 15-months
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | mPEP | Bibliotherapy
Number analyzed (Participants) | 63 | 52
Scores on a scale
  Positive Affect | 30.0 (0.97) | 29.8 (0.98)
  Negative Affect | 20.4 (0.95) | 19.5 (0.98)

3. Secondary Outcome: Blood Pressure
Description: Systolic and Diastolic Blood Pressure
Time Frame: 15-months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | mPEP | Bibliotherapy
Number analyzed (Participants) | 63 | 52
mmHg
  Systolic Blood Pressure | 123.4 (2.1) | 121.3 (1.9)
  Diastolic Blood Pressure | 75.8 (1.2) | 76.0 (1.3)

4. Secondary Outcome: Dementia Quality of Life Scale for Older Family Carers (DQoLOC)
Description: Dementia Quality of Life Scale for Older Family Carers (DQoLOC). Scale consists of 22 items, each item is rated from 1-5. The total range for the scale is 22-110, with higher score indicating greater quality of life.
Time Frame: 15-months
Population: Participant withdrawal and lost to follow-up
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | mPEP | Bibliotherapy
Number analyzed (Participants) | 63 | 52
Score on a scale | 63.5 (1.9) | 64.8 (2.0)

ADVERSE EVENTS:
Time Frame: From enrollment until 15 months
Description: Clinical Trials definitions
Arm/Group | mPEP | Bibliotherapy
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/91
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/91
Other Adverse Events (participants affected / at risk) | 12/93 | 13/91
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mPEP (N=93) | Bibliotherapy (N=91)
Progression of Dementia (General disorders) | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03506945/Prot_SAP_000.pdf